CLINICAL TRIAL: NCT00097422
Title: An Open-Label, Dose Ranging, Randomized Clinical Evaluation of OPT-80 in Patients With Clostridium Difficile-Associated Diarrhea (CDAD)
Brief Title: OPT-80 in Clostridium Difficile-Associated Diarrhea (CDAD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Optimer Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5119-022; OPT-80 Phase 2A (Other: Optimerpharma Study Number)
Record Dates: First submitted 2004-11-23; First posted 2004-11-24 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Diarrhea
Keywords: CDAD, diarrhea; Clostridium difficile-Associated Diarrhea
MeSH Terms: conditions — Diarrhea | interventions — OPT 80

INTERVENTIONS:
Drug: OPT-80

SUMMARY:
The purpose of this study is to investigate the safety and perform preliminary clinical evaluation in patients with mild to moderate CDAD.

DETAILED DESCRIPTION:
This is a dose-finding study to select a safe and efficacious dose of OPT-80. Patients will be evaluated for safety and efficacy and pharmacokinetic parameters will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CDAD

Exclusion Criteria:

* Patients with severe CDAD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-11-01 (Actual); Primary Completion 2005-04-01 (Actual); Study Completion 2005-04-01 (Actual)

PRIMARY OUTCOMES:
Relief of symptoms of CDAD

SECONDARY OUTCOMES:
Recurrence Rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Biologics, New Hope, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Louie T, Miller M, Donskey C, Mullane K, Goldstein EJ. Clinical outcomes, safety, and pharmacokinetics of OPT-80 in a phase 2 trial with patients with Clostridium difficile infection. Antimicrob Agents Chemother. 2009 Jan;53(1):223-8. doi: 10.1128/AAC.01442-07. Epub 2008 Oct 27. PMID 18955525